CLINICAL TRIAL: NCT05430191
Title: Leveraging Behavioral Economics to Equitably Implement Cascade Screening in Individuals With Familial Hypercholesterolemia in Partnership With the Family Heart Foundation
Brief Title: Equitable Implementation of Cascade Screening for Familial Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Family Heart Foundation (Unknown); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Rinad Beidas, Ralph Seal Paffenbarger Professor and Chair, Department of Medical Social Sciences, Northwestern University
Other Study IDs: 851061
Record Dates: First submitted 2022-06-08; First posted 2022-06-24 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Qualitative Interviews: Conduct 15 interviews with patients diagnosed with FH. Interviews will be 30-60 minutes in length and will focus on how individuals understand cascade screening, barriers to engagement including reasons why individuals do and do not share health information with family members, and preferred approaches to engaging family members, with a focus on acceptability, appropriateness, and feasibility of the planned implementation strategies. Interviewers will also attend to structural factors such as medical mistrust and experiences of racism in health care, and ask about preferences and logistics to incorporate preference into the future clinical trial design.
- Penn-mediated implementation strategy: The Penn-mediated implementation strategy will be designed and then iterated upon during mini-pilots. As part of this strategy, the patients would receive text messages and/or emails containing information about FH and cascade screening from Penn Medicine. This would include a request for the patient to identify first-degree biological relatives. They would be given a choice of either contacting their family members directly or sharing their contact information so someone from Penn Medicine can contact them. If the proband chooses to contact their family members, they receive educational information to share with them. Family members would be offered FH screening at no cost by blood lipid panel.
  Interventions: Other: Cascade Screening
- Family Heart Foundation-mediated implementation strategy: The Family Heart Foundation (FHF)-mediated implementation strategy will be designed and then iterated upon during mini-pilots. As part of this strategy, the patient would be contacted by a FHF patient navigator. The patient navigator would ask to set up a time to talk to the patient to talk about options for contacting family members, introduce them to the services they can provide to the patient and/or family members and obtain some details about the patient's family. The patient would come up with a plan to either contact their family members directly or have the patient navigator contact them. Family members will be offered FH screening at no cost by blood lipid panel. The patient and/or family members will be able to contact the patient navigator at any time with questions.
  Interventions: Other: Cascade Screening

INTERVENTIONS:
Other: Cascade Screening — FH is a genetic condition that causes high LDL cholesterol starting at birth. When one individual with FH is diagnosed, it is important that biological family members are also screened, since there is a 50% chance that each first-degree relative will have also inherited FH. More distant relatives may also have inherited FH. This evidence-based process is known as cascade screening.
  Groups: Family Heart Foundation-mediated implementation strategy; Penn-mediated implementation strategy

SUMMARY:
Design, refine, and pilot the two implementation approaches using behavioral economics and then seek further feedback prior to the proposed clinical trial, consistent with these recommendations.

Aim 1. Co-design both implementation strategies using behavioral economics in partnership with the Family Heart Foundation and key partners from diverse backgrounds.

Aim 2. Pilot strategies with 20 patients with high cholesterol and/or with familial hypercholesterolemia (FH) to ascertain feasibility, acceptability, appropriateness.

DETAILED DESCRIPTION:
Aim 1. Conduct interviews with patients with high cholesterol and/or FH and clinicians to identify common barriers and facilitators for individuals to engage in cascade screening. These activities will occur in the first 7 months and will serve as inputs into the design of the implementation strategies to ensure that strategies address determinants identified in the interviews.

Aim 2. To maximize success, pilot test the implementation strategies and the planned data collection approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high cholesterol and/or FH (i.e., probands; Aim 1 Interviews, Aim 2 Pilot Testing Strategies, Aim 2 Interviews). Adults aged 18 and older with clinically diagnosed FH and/or high cholesterol who are treated within Penn Medicine.
* Family Members (Aim 2 Pilot Testing Strategies, Aim 2 Interviews). Adults aged 18 and older who have a family member who has been identified as a patient with high cholesterol and/or FH who is treated within Penn Medicine (i.e., family members of probands).

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aim 1 (Interviews). We will conduct interviews with 15 patients with high cholesterol and/or FH to understand barriers and facilitators to cascade screening. 17 clinicians are being interviewed through our sister protocol in an effort to reduce interview burden on clinicians. Duration of participation will last the length of one qualitative interview.
  Aim 2 (Pilot Testing Strategies). Participants will include 20 patients with high cholesterol and/or FH. At least half will identify as racial and/or ethnic minorities (i.e., Black or African American, Asian), female, and/or have low income. Patients will be randomized to receive the Penn- or FHF-mediated strategy. Duration of participation will last up to 3 months for each participant.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Aim 1 Qualitative Interview Outcome: Perspectives on cascade screening | 1-time interview to last 1 hour
  We will learn about the perspectives on cascade screening from clinicians and patients with high cholesterol and/or FH (probands) via qualitative interview.
Aim 2 Mini-Pilot Outcome: Engagement | 3 months
  We define engagement as the number of patients with FH and/or high cholesterol (probands) who respond to at least one outreach attempt.
Aim 2 Mini-Pilot Outcome: Reach | 3 months
  We define reach as the proportion of probands who have at least one family member who completes cascade screening.
Aim 2 Mini-Pilot Outcome: Perspectives on implementation strategies | 1-time interview to last approximately 15-30 minutes
  We will learn about the perspectives on the implementation strategies (health system-mediated, Family Heart Foundation-mediated) - including their perceived acceptability, appropriateness, and feasibility - of patients with high cholesterol and/or FH (probands) and family members via qualitative interview.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT05430191/Prot_SAP_002.pdf
  • Informed Consent Form: Aim 2 (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT05430191/ICF_003.pdf
  • Informed Consent Form: Aim 1 (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT05430191/ICF_004.pdf